CLINICAL TRIAL: NCT01615809
Title: A Phase II Trial to Evaluate the Safety and Tolerability of Nebulised Amphotericin B Lipid Complex (ABELCET®) in the Prophylaxis of Invasive Pulmonary Aspergillosis During Prolonged Neutropenia in Paediatric Patients With Acute Leukaemia
Brief Title: Nebulized Amphotericin B Lipid Complex in Invasive Pulmonary Aspergillosis in Paediatric Patients With Acute Leukaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSJD-ABELNEB-2010
Record Dates: First submitted 2012-06-04; First posted 2012-06-11 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Invasive Pulmonary Aspergillosis; Lymphoblastic Leukaemia; Myeloblastic Leukaemia; Lymphoblastic Leukemia; Myeloblastic Leukemia
Keywords: Invasive pulmonary aspergillosis; IFI; Leukaemia; Leukemia; Pediatric; Paediatrics; Amphotericin B; Aspergillosis; Pulmonary Aspergillosis; Invasive Aspergillosis; Antifungal agents; Fungal infections; Invasive Fungal Infection
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Acute; Leukemia; Aspergillosis; Pulmonary Aspergillosis; Mycoses; Invasive Fungal Infections | interventions — Amphotericin B; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amphotericin B (ABELCET®) (Experimental): Drug: AMPHOTERICIN B Dosage form: Abelcet® 5mg/ml administered by inhalation. Dosage: 10 ml (50 mg) for the first week with a frequency twice a week. Dosage: from the second week onwards 5 ml (25 mg) with a frequency of a minimum separation of 72 hours between doses, until the neutrophil count is greater than or equal to 1500 cells/mm3.
  Duration: 4-5 prophylaxis courses defined as each administration period during a neutropenia period, with a 4-6 weeks length considering the duration of neutropenia.
  Interventions: Drug: AMPHOTERICIN B

INTERVENTIONS:
Drug: AMPHOTERICIN B — The study drug will be administered by inhalation, to hospitalised patients or outpatients in the day hospital.
  Other Names: Abelcet® 5 mg/ml

SUMMARY:
The trial evaluates the overall tolerability of the drug and the efficacy of aerosolised amphotericin B as a lipid complex (ABLC) for primary prophylaxis of invasive pulmonary aspergillosis (IPA) in pediatric patients with acute leukemia undergoing intensive chemotherapy.

DETAILED DESCRIPTION:
In recent years the incidence of invasive fungal infection (IFI) especially when caused by filamentous fungi has increased in patients with haematological malignancies and there exists an international consensus on diagnostic criteria. Despite diagnostic and therapeutic progress, invasive aspergillosis remains a major clinical problem of haematological patients, given the still high mortality rates and the huge economic cost of hospitalization of patients, which is attributable to aspergillosis. In addition to the morbidity and mortality rates, these infections interfere with the chemotherapy treatment plan with the risk of compromising the outcome of the antileukemic treatment.

In a few uncontrolled studies inhaled amphotericin B deoxycholate showed some benefit in haematological patients, however it was not effective in a large multicenter study with neutropenic patients. Based on the outcome of that clinical trial, the use of aerosolised amphotericin B deoxycholate in neutropenic patients was abandoned for nearly a decade. During this time the use of azole agents as drugs of choice for antifungal prophylaxis in high risk patients was consolidated. However, one of the main problems in the use of triazoles with activity against filamentous fungi (itraconazole, voriconazole, posaconazole) is drug-drug interactions due to their CYP3A4 inhibitory activity. One of the most serious interactions is that which occurs with vincristine, used throughout the treatment of acute lymphoblastic leukemia, and which has lead to reports of neurotoxicity due to metabolic inhibition.

ABLC (Abelcet®) belongs to the group of polyenes with antifungal activity against a broad spectrum of fungal species, including Aspergillus spp. The active component of ABELCET®, amphotericin B, acts by binding to sterols in the cell membrane of susceptible fungi, with a resultant change in the permeability of the membrane. Mammalian cell membranes also contain sterols, and damage to human cells is believed to occur through the same mechanism of action.

Abelcet® is recommended for the intravenous treatment of a broad spectrum of systemic fungal infections in adult patients. Although it has a pediatric indication, there are numerous studies published regarding the safety levels of Abelcet® administered intravenously in children and in haematological adults patients which look very promising. In this context, the working hypothesis proposed in this project is that the administration of aerosolised ABLC for pediatric patients with acute leukemia treated with intensive chemotherapy will be an effective alternative as a prophylaxis of pulmonary fungal infections in these patients.

In the treatment of pediatric patients with haematological malignancies the use of intensive chemotherapy is required, which is immunosuppressive and therefore significantly increases the risk of IFI, especially filamentous fungi. IPA is associated with high mortality (>50%) in those patients, making it imperative to adopt effective, preventive, prophylactic measures. Drug interactions occur frequently with triazole antifungal drugs; cases of clinically significant interactions with vincristine, an anchor drug in the treatment of the majority of pediatric leukemia, are documented. On the other hand, there are promising data from previous studies regarding the safety and efficacy of the intravenous ABLC formulation (Abelcet®) in the treatment of pediatric patients with fungal infections.

If the working hypothesis is confirmed, the aerosolised ABLC treatment would be an effective, safe and reliable prophylactic option for IPA. It would offer an alternative to the systemic administration of antifungal triazoles without affecting the antileukemic treatment in pediatric patients with AL.

ELIGIBILITY:
Inclusion Criteria:

1. Age: patients between 3 and 18 years.
2. Diagnosis of myeloblastic or lymphoblastic AL during intensive chemotherapy.
3. Informed consent of parents/guardians and/or assent of the patient has been obtained.

Exclusion Criteria:

1. Probable or proven invasive pulmonary fungal infection before entering the trial.
2. Previous chronic renal impairment or baseline serum creatinine > 2.5 mg /dL
3. Severe hepatic impairment.
4. Moderate-severe asthma being treated pharmacologically.
5. Antifungal treatment for filamentous fungi in the last 4 weeks.
6. Participating or have participated in a clinical trial during the last 4 weeks.
7. Mentally retarded
8. Known allergy or hypersensitivity to the active ingredient of the study drug or to any of its excipients.
9. Any serious concomitant disease that in the investigator's opinion could compromise the completion of the trial or affect the patient's tolerability to this treatment.
10. Pregnancy (in women of fertile age).
11. Breast-feeding.

Patients are defined as having probable IFI when their radiological image is suggestive of fungal infection and they have positive antigenemia for Aspergillus. IFI would be proven when the presence of Aspergillus is confirmed in aspirate culture or by lung biopsy.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Estella, PhMD, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data of participants will be shared with Authorities at the end of the Clinical Development Plan by the CTD (Common Technical Document). Results will be published in a scientific publication.

REFERENCES:
- [Background] Ascioglu S, Rex JH, de Pauw B, Bennett JE, Bille J, Crokaert F, Denning DW, Donnelly JP, Edwards JE, Erjavec Z, Fiere D, Lortholary O, Maertens J, Meis JF, Patterson TF, Ritter J, Selleslag D, Shah PM, Stevens DA, Walsh TJ; Invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer; Mycoses Study Group of the National Institute of Allergy and Infectious Diseases. Defining opportunistic invasive fungal infections in immunocompromised patients with cancer and hematopoietic stem cell transplants: an international consensus. Clin Infect Dis. 2002 Jan 1;34(1):7-14. doi: 10.1086/323335. Epub 2001 Nov 26. PMID 11731939
- [Background] Walsh TJ, Gonzalez C, Lyman CA, Chanock SJ, Pizzo PA. Invasive fungal infections in children: recent advances in diagnosis and treatment. Adv Pediatr Infect Dis. 1996;11:187-290. No abstract available. PMID 8718464
- [Background] Blyth CC, Palasanthiran P, O'Brien TA. Antifungal therapy in children with invasive fungal infections: a systematic review. Pediatrics. 2007 Apr;119(4):772-84. doi: 10.1542/peds.2006-2931. PMID 17403849
- [Background] Bodey GP, Anaissie EJ, Elting LS, Estey E, O'Brien S, Kantarjian H. Antifungal prophylaxis during remission induction therapy for acute leukemia fluconazole versus intravenous amphotericin B. Cancer. 1994 Apr 15;73(8):2099-106. doi: 10.1002/1097-0142(19940415)73:83.0.co;2-n. PMID 8156515
- [Background] Lin SJ, Schranz J, Teutsch SM. Aspergillosis case-fatality rate: systematic review of the literature. Clin Infect Dis. 2001 Feb 1;32(3):358-66. doi: 10.1086/318483. Epub 2001 Jan 26. PMID 11170942
- [Background] Perfect JR, Klotman ME, Gilbert CC, Crawford DD, Rosner GL, Wright KA, Peters WP. Prophylactic intravenous amphotericin B in neutropenic autologous bone marrow transplant recipients. J Infect Dis. 1992 May;165(5):891-7. doi: 10.1093/infdis/165.5.891. PMID 1569339
- [Background] Walsh TJ, Hiemenz J, Pizzo PA. Evolving risk factors for invasive fungal infections--all neutropenic patients are not the same. Clin Infect Dis. 1994 May;18(5):793-8. doi: 10.1093/clinids/18.5.793. No abstract available. PMID 8075273
- [Background] Walsh TJ, Hiemenz JW, Anaissie E. Recent progress and current problems in treatment of invasive fungal infections in neutropenic patients. Infect Dis Clin North Am. 1996 Jun;10(2):365-400. doi: 10.1016/s0891-5520(05)70303-2. PMID 8803625
- [Background] Walsh TJ, Finberg RW, Arndt C, Hiemenz J, Schwartz C, Bodensteiner D, Pappas P, Seibel N, Greenberg RN, Dummer S, Schuster M, Holcenberg JS. Liposomal amphotericin B for empirical therapy in patients with persistent fever and neutropenia. National Institute of Allergy and Infectious Diseases Mycoses Study Group. N Engl J Med. 1999 Mar 11;340(10):764-71. doi: 10.1056/NEJM199903113401004. PMID 10072411
- [Background] Herbrecht R. The changing epidemiology of fungal infections: are the lipid-forms of amphotericin B an advance? Eur J Haematol Suppl. 1996;57:12-7. doi: 10.1111/j.1600-0609.1996.tb01347.x. PMID 8706811
- [Background] Herbrecht R. Improving the outcome of invasive aspergillosis: new diagnostic tools and new therapeutic strategies. Ann Hematol. 2002;81 Suppl 2:S52-3. No abstract available. PMID 12611078
- [Background] Nakagawa Y. [Prophylactic administration of fluconazole and itraconazole in febrile neutropenia associated with hematopoietic malignancy]. Jpn J Antibiot. 2006 Oct;59(5):407-9. No abstract available. Japanese. PMID 17205660
- [Background] Boettcher H, Bewig B, Hirt SW, Moller F, Cremer J. Topical amphotericin B application in severe bronchial aspergillosis after lung transplantation: report of experiences in 3 cases. J Heart Lung Transplant. 2000 Dec;19(12):1224-7. doi: 10.1016/s1053-2498(00)00154-6. PMID 11124494
- [Background] Alexander BD, Dodds Ashley ES, Addison RM, Alspaugh JA, Chao NJ, Perfect JR. Non-comparative evaluation of the safety of aerosolized amphotericin B lipid complex in patients undergoing allogeneic hematopoietic stem cell transplantation. Transpl Infect Dis. 2006 Mar;8(1):13-20. doi: 10.1111/j.1399-3062.2006.00125.x. PMID 16623816
- [Background] Rijnders BJ, Cornelissen JJ, Slobbe L, Becker MJ, Doorduijn JK, Hop WC, Ruijgrok EJ, Lowenberg B, Vulto A, Lugtenburg PJ, de Marie S. Aerosolized liposomal amphotericin B for the prevention of invasive pulmonary aspergillosis during prolonged neutropenia: a randomized, placebo-controlled trial. Clin Infect Dis. 2008 May 1;46(9):1401-8. doi: 10.1086/586739. PMID 18419443

RESULTS

PARTICIPANT FLOW:
Groups:
- Amphotericin B (ABELCET®): Patients fulfilling inclusion criteria and those giving the general informed consent for the study will initiate nebulized Amphotericin B prophylaxis treatment, twice a week, during neutropenia periods (coincident with intensive chemotherapy treatment).
  AMPHOTERICIN B: The study drug will be administered by inhalation, to hospitalised patients or outpatients in the day hospital.The administration regimen for each Abelcet® nebulization will be 10 ml (50 mg) twice a week for the first week, and then from the second week onwards it will be 5 ml (25 mg) with a minimum separation of 72 hours between doses, until the neutrophil count is greater than or equal to 1500 cells/mm3.
Period: Overall Study
Arm/Group | Amphotericin B (ABELCET®)
Started | 32 (basal visit)
Completed | 22
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: pediatric patients
Groups:
- Amphotericin B (ABELCET®): Patients fulfilling inclusion criteria and those giving the general informed consent for the study initiate nebulized Amphotericin B prophylaxis treatment, twice a week, during neutropenia periods (coincident with intensive chemotherapy treatment).
  AMPHOTERICIN B: The study drug will be administered by inhalation, to hospitalised patients or outpatients in the day hospital.The administration regimen for each Abelcet® nebulization was 10 ml (50 mg) twice a week for the first week, and then from the second week onwards was reduced to 5 ml (25 mg) with a minimum separation of 72 hours between doses, until the neutrophil count demonstrated to be greater than or equal to 1500 cells/mm3.
Arm/Group | Amphotericin B (ABELCET®)
Number analyzed (Participants) | 32
Age, Customized [Number; unit: participants]
  >= 3 years to <=18 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants] — patients ethnicity percentage : caucasian (84.4%), Amerindian (6.3%), African (3.1%) and gypsies (6.3%).
  participants
    caucasian | 27
    amerindian | 2
    african | 1
    gypsies | 2
Region of Enrollment [Number; unit: center]
  Spain | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events That Results in the Interruption of Treatment, as a Measure of Safety and Tolerability
Description: is assessed by the proportion of patients who discontinue prophylactic treatment with Abelcet® due to an adverse event that is related or not to the study drug or for intolerability to it. The last week of treatment will have a different calendar for each participant, depending on the number of cicles needed by each patient (it has been anticipated up to 5 cicles of 2-6 weeks each).
Time Frame: at the Baseline visit (week 1) and during the Last week of treatment, up to 6 weeks
Population: pediatric patients
Measure: Number; unit: participants
Arm/Group | Amphotericin B (ABELCET®)
Number analyzed (Participants) | 32
participants | 0

2. Secondary Outcome: Efficacy of Primary Prophylaxis With Nebulized Abelcet® on the Incidence of Invasive Pulmonary Aspergillosis
Description: The incidence of invasive pulmonary aspergillosis during the Abelcet® prophylactic treatment period was assessed by the relation between the number of patients with invasive pulmonary aspergillosis and the number of paediatric patients on prophylaxis with Acute Leukaemia (AL) undergoing intensive chemotherapy.
Time Frame: at the Baseline visit (week 1) and at the end of the profilaxis treatment phase, up to 6 weeks
Population: At baseline, none of the 32 pediatric patients with acute leukemia included in the clinical trial had API. During the trial period there were 3 patients who developed API
Measure: Number; unit: participants
Arm/Group | Amphotericin B (ABELCET®)
Number analyzed (Participants) | 32
participants | 3

3. Secondary Outcome: Invasive Pulmonary Aspergillosis -Related Mortality During Primary Prophylaxis With Abelcet®.
Description: Percentage of deaths related to Invasive Pulmonary Aspergillosis during the prophylactic treatment period with Abelcet® in paediatric patients with Acute Leukaemia undergoing intensive chemotherapy.
Time Frame: at the Baseline visit (week 1) and at the end of the profilaxis treatment phase, up to 6 weeks
Measure: Number (95% Confidence Interval); unit: percentage of deaths
Arm/Group | Amphotericin B (ABELCET®)
Number analyzed (Participants) | 32
percentage of deaths | 0 [0 to 0]

ADVERSE EVENTS:
Arm/Group | Amphotericin B (ABELCET®)
Serious Adverse Events (participants affected / at risk) | 22/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amphotericin B (ABELCET®) (N=32)
febrile neutropenia (Blood and lymphatic system disorders) | 16 (26)
fever (General disorders) | 8 (13)
hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Febrile Aplasia (Blood and lymphatic system disorders) | 3 (3)
Methotrexate-induced neurotoxicity (Nervous system disorders) | 3 (3)
macroscopic hematuria (Blood and lymphatic system disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amphotericin B (ABELCET®) (N=32)
Fever (General disorders) | 32 (32)
abdominal pain (Gastrointestinal disorders) | 29 (32)
paleness (General disorders) | 28 (32)
physical pain (General disorders) | 24 (32)
diarrhea (Gastrointestinal disorders) | 21 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days